CLINICAL TRIAL: NCT03328741
Title: Evaluation of a Web-based Platform for Osteoarthritis Treatment - a Randomized Clinical Trial
Brief Title: Evaluation of a Web-based Platform for Osteoarthritis Treatment
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OA-treatment RCT
Record Dates: First submitted 2017-09-22; First posted 2017-11-01 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Osteoarthritis, Knee
Keywords: Clinical Trials, Randomized; Telemedicine
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Joint Academy (Experimental): Online osteoarthritis treatment
  Interventions: Behavioral: Online Osteoarthritis treatment
- The BOA program (Active Comparator): Face-to-face osteoarthritis treatment
  Interventions: Behavioral: Face-to-face osteoarthritis treatment

INTERVENTIONS:
Behavioral: Online Osteoarthritis treatment — 6 week online-program
  Other Names: Joint Academy
  Arms: Joint Academy
Behavioral: Face-to-face osteoarthritis treatment — 3 months face-to-face program
  Other Names: The BOA program
  Arms: The BOA program

SUMMARY:
This study will compare the effects of a novel web-based program (Joint Academy) to regular face-to-face treatment (the BOA program) for people with osteoarthritis of the knee. Half of the participants will be randomized to the web-based program whilst the other half will receive regular face-to-face care.

DETAILED DESCRIPTION:
According to national and international guidelines, osteoarthritis (OA) treatment consists of exercise and information. The face-to-face BOA program is a model to deliver this treatment at primary care facilities in Sweden. Presently less than 20% of people with OA receive adequate treatment. This may be due to lack of healthcare resources or people having trouble to fit their schedule to primary care opening hours. To facilitate a better OA care, alternative methods are therefore required.

A two-armed randomized clinical superiority trial will be performed to compare OA treatment by a web-based program, Joint Academy, with the traditional face-to-face BOA program in 270 adults with clinically verified OA. Using intention-to-treat analysis and per-protocol, evaluations will be performed at baseline, after 6 weeks and after 3, 6 and 12 months. The primary outcome is physical function. Secondary outcomes are joint pain, health-related quality of life, self-reported function, amount of time of physical activity/exercise and overall satisfaction. A health-economic analysis will also be performed. The primary endpoint will be at 12 months. Data will be monitored using web-based questionnaires in Joint Academy, and regular paper questionnaires for the face-to-face treatment.

Should the trial show superiority in favor of Joint Academy, an implementation of the web-based treatment would benefit both patient and society at large, since Joint Academy entails a more flexible treatment in regards to time and location, and is not as costly per-patient as regular face-to-face treatment.

ELIGIBILITY:
Inclusion criteria:

I: A clinical diagnosis of knee OA according to American College of Rheumatology (ACR) diagnostic criteria as well as national and international guidelines: knee pain and 3 of the following: > 50 years of age, morning stiffness >30 min, crepitus, bony tenderness, bony enlargement, no palpable warmth; II: Reported knee pain ≥4 and ≤8 on the NRS, and ≥6 to ≤16 in number of repetitions of the 30 second chair stand test, at pre-randomization screening.

II: Able to handle a software program via phone, tablet or computer. III: Able to read and write the Swedish language.

Exclusion criteria:

I: Neurological disease, inflammatory joint disease or cancer. II: Cognitive disorder, e.g. dementia. III: Exercise is contra-indicated for the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2018-05-22 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Physical functioning | Change from baseline to 6 months (3 months after end of treatment) and at 12 month follow-up
  Measured using the 30 second chair stand test, defined in number of repetitions. The result is directly reported after test performance

SECONDARY OUTCOMES:
NRS pain | Change from baseline to 6 months (3 months after end of treatment) and at 12 month follow-up
  Self-reported knee pain on a 0-10 numeric rating scale (NRS) reported as during the latest week
Health-related quality of life | Change from baseline to 6 months (3 months after end of treatment) and at 12 month follow-up
  Measured using the EQ5D-5L, index value. Measures the patients status at the day of reporting
Self-reported function | Change from baseline to 6 months (3 months after end of treatment) and at 12 month follow-up
  Measured using the KOOS-ps, for the latest week.
Physical activity | Change from baseline to 6 months (3 months after end of treatment) and at 12 month follow-up
  Number of minutes of physical activity and exercise per week.

CONTACTS AND LOCATIONS:
Overall Officials: Håkan Nero, PhD, Principal Investigator — Department of Orthopaedics, Lund University
Locations (1):
- Abels Rehab, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD for primary and secondary outcomes will be made available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Study protocol, SAP and ICF will be made available six months after study completion. CSR and Analytic Code will be available after publication of results.
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Derived] Nero H, Ranstam J, Kiadaliri AA, Dahlberg LE. Evaluation of a digital platform for osteoarthritis treatment: study protocol for a randomised clinical study. BMJ Open. 2018 Nov 8;8(11):e022925. doi: 10.1136/bmjopen-2018-022925. PMID 30413507